CLINICAL TRIAL: NCT06884982
Title: An Exploratory Clinical Study on Neoadjuvant Treatment of Hepatocellular Carcinoma with Iparomlimab and Tuvonralimab Injection Combined with Lenvatinib
Brief Title: An Exploratory Clinical Study on Neoadjuvant Treatment of Hepatocellular Carcinoma with QL1706 Combined with Lenvatinib
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025ky032
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: HCC - Hepatocellular Carcinoma
Keywords: neoadjuvant therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- QL1706 plus lenvatinib (Experimental)
  Interventions: Drug: QL1706 Plus Lenvatinib

INTERVENTIONS:
Drug: QL1706 Plus Lenvatinib — All enrolled subjects will receive QL1706 5 mg/kg intravenously plus lenvatinib 8/12mg on day 1 of each cycle (every 3 weeks). Tumor assessment will be done after 6 weeks (2 cycles) and 12 weeks (4 cycles).

SUMMARY:
This is a single-center, single-arm, prospective trial to explore the efficacy and safety of neoadjuvant treatment with Iparomlimab and Tuvonralimab Injection combined with lenvatinib in patients with advanced HCC

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤ 75 years；
2. Confirmed by pathological or imaging diagnosis as CNLC Ib/IIa/IIb/IIIa HCC (fibrotic plate and mixed hepatocellular/cholangiocarcinoma subtypes do not meet the inclusion criteria);
3. Patients who have not received surgery or systemic treatment before enrollment and have experienced recurrence within 2 years after surgery can be included;
4. MDT team determines that HCC with high-risk factors for recurrence (such as macroscopic cancer thrombus, multiple tumors, satellite nodules, tumor diameter > 5 cm, imaging vascular invasion or preoperative AFP > 200 U/ml) is resectable;
5. Positive hepatitis B surface antigen, no restrictions on anti-hepatitis B virus treatment;
6. At least one measurable lesion based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) evaluated by the investigator;
7. Organ function levels must meet the following requirements: i. Adequate bone marrow reserve: absolute neutrophil count >= 1.5 x 10^9/L, white blood cell count >= 3 x 10^9/L, platelet count >= 90 x 10^9/L, and hemoglobin >= 9 g/dL; ii. Liver: plasma albumin >= 2.8 g/dL; for patients without liver metastasis, serum bilirubin <= 2xULN, and for patients with liver metastasis, serum bilirubin <= 3xULN; for patients without liver metastasis, AST and ALT <= 2.5xULN, and for patients with liver metastasis, AST and ALT <= 5xULN; iii. Kidney: serum creatinine <= 1.5xULN; iv. Heart: left ventricular ejection fraction (LVEF) >= 50% (no blood transfusion, no use of hematopoietic growth factors and human albumin within 14 days before screening);
8. Non-surgical sterilized female or male subjects of childbearing age, must agree to use a medically approved contraceptive method (such as intrauterine device, contraceptive pills or condoms) for contraception during the study treatment period and within 6 months after the end of the study treatment period; for non-surgical sterilized female subjects, the HCG test must be negative within 7 days before enrollment and must not be lactating;
9. Child-Pugh: A/B grade (<= 7 points);
10. ECOG performance status 0-1;
11. Expected survival >= 6 months.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Patients with imaging evidence showing portal vein tumor thrombus reaching Vp3 or Vp4;
3. Patients who have received PD-1 antibody, PD-L1 antibody, CTLA-4 antibody or lenvatinib before; those who participated in other clinical trials within 30 days before screening;
4. Patients with active tuberculosis infection. Those who have active pulmonary tuberculosis within 1 year before enrollment; those who have had active tuberculosis infection for more than 1 year before enrollment and have not received regular anti-tuberculosis treatment or tuberculosis is still active;
5. Patients with gastrointestinal malabsorption, gastrointestinal anastomosis or any other conditions that may affect the absorption of lenvatinib;
6. Patients with NYHA II grade or above congestive heart failure history, unstable angina pectoris, myocardial infarction within 6 months or severe arrhythmia with significant cardiovascular damage within 6 months;
7. Within 3 weeks before the first administration of the study drug, patients have experienced gastrointestinal bleeding events or active hemoptysis (at least 0.5 teaspoons of bright red blood);
8. Patients with bleeding or thrombotic diseases or using X-factor inhibitors or anticoagulants that require monitoring of the international normalized ratio (INR), such as warfarin or similar drugs. Low molecular weight heparin treatment is allowed. Antiplatelet drugs at the treatment dose (such as aspirin ≥ 325 mg/d) are not allowed to be used during the study process;
9. Patients who require immunosuppressive therapy after organ transplantation; patients who have received immunosuppressive drugs or systemic corticosteroids to achieve immunosuppression purposes within 14 days before enrollment (such as > 10 mg/day prednisone or equivalent drugs);
10. Patients with active ulcers, unhealed wounds or fractures;
11. Patients with hypertension and poor control of blood pressure (systolic blood pressure >= 140 mmHg or diastolic blood pressure >= 90 mmHg);
12. Patients known to be allergic to any trial drug or excipients;
13. Patients who have had other malignant tumors that have not been cured for more than 5 years, but do not include clearly cured malignant tumors, or curable cancers, such as basal cell carcinoma or squamous cell carcinoma of the skin, papillary thyroid carcinoma, localized low-risk prostate cancer, cervical carcinoma in situ or breast carcinoma in situ, etc.;
14. Patients who have received allogeneic tissue/organ transplantation;
15. Patients with known HIV infection history;
16. According to the investigator's judgment, the subjects have other factors that may affect the trial results or cause the study to be forced to stop prematurely, such as alcohol abuse, drug abuse, other serious diseases (including mental diseases) that require combined treatment, severe laboratory test abnormalities, and factors affecting the patient's safety due to family or social factors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-13 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who obtain a major pathologic responses (MPR) | 3 years

SECONDARY OUTCOMES:
Percentage of participants who obtain a pathologic complete response (CR). | 4 years
Percentage of participants who obtain R0 resection. | 4 years
Event-Free Survival(EFS) | 4 years

IPD SHARING:
Plan to Share IPD: No